CLINICAL TRIAL: NCT01229982
Title: A Phase 2 Study Evaluating Safety and Efficacy of the Latanoprost Punctal Plug Delivery System (L PPDS)in Subjects With Ocular Hypertension (OH) or Open Angle Glaucoma (OAG)
Brief Title: A Study Evaluating the Latanoprost Punctal Plug Delivery System (L-PPDS) in Subjects With Ocular Hypertension or Open-Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPL GLAU 11
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-PPDS (Experimental)
  Interventions: Drug: Latanoprost-PPDS

INTERVENTIONS:
Drug: Latanoprost-PPDS — Punctal Plug

SUMMARY:
The purpose of this study is to test if latanoprost punctal plugs will reduce eye pressure in subjects with ocular hypertension or open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bilateral OH or OAG and on topical prostaglandin monotherapy bilaterally as standard of care for treatment of OH or OAG.
* Adequate IOP control on topical prostaglandin monotherapy during the past 1 month.

Exclusion Criteria:

* Functionally significant vision loss, or progressive field loss within the last year.
* Contact lens wear at any time during the treatment period.
* Keratoconjunctivitis sicca requiring chronic topical artificial tears, lubricants, and/or Restasis®.
* Active lid disease (i.e., moderate or severe blepharitis, meibomianitis) that requires medical treatment.
* Subjects with ≥0.9 vertical cup or completely notched optic nerve head rim.
* Currently on chronic ocular topical medications
* Currently on any ophthalmic or systemic steroid therapy.
* Laser surgery for glaucoma within the last 3 months or 6 months for incisional surgeries.
* History of macular edema
* History of chronic/recurrent inflammatory eye disease.
* History of a non-response to topical prostaglandin therapy.
* Subjects who have epiphora.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
IOP change from baseline at 4 weeks | Baseline to 4 Weeks
  4 Weeks minus baseline

CONTACTS AND LOCATIONS:
Locations (1):
- QLT Inc., Vancouver, British Columbia, Canada